CLINICAL TRIAL: NCT06641193
Title: A Randomized Sham-Controlled Trial of High-frequency RTMS in the Treatment of Upper Limb Bradykinesia in Patients with Parkinson's Disease
Brief Title: Clinical Trail of Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Upper Limb Bradykinesia in Parkinson' Disease' Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhengguo Liu, Director of Department of Neurology, Principal Investigator, Clinical Professor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XHEC-C-2024-125-2-2
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-08

CONDITIONS: Parkinson's Disease (PD); Bradykinesia; Upper Limb Function
MeSH Terms: conditions — Hypokinesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- verum group (Experimental): verum group receive real 10 sessions of rTMS stimulation. once daily for 5 consecutive days a week.
  Interventions: Device: high frequency-repetitive transcranial magnetic stimulation
- sham group (Sham Comparator): The sham group receives 10 sessions of rTMS stimulation, once daily for 5 consecutive days a week. However, a sham stimulation coil is used, which emits the same sound and vibration as the active coil but does not produce any induced electrical currents.
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: high frequency-repetitive transcranial magnetic stimulation — rTMS involves the repeated application of magnetic pulses to specific areas of the brain. These pulses are delivered using a coil placed on the scalp, which generates a magnetic field that induces electrical currents in the brain tissue.
  Arms: verum group
Device: sham stimulation — The sham group receives 10 sessions of rTMS stimulation with a sham stimulation coil, which emits the same sound and vibration as the active coil but does not produce any induced electrical currents.
  Arms: sham group

SUMMARY:
A randomized, double-blind, sham-controlled unicenter clinical trial was used to investigate the effectiveness and neural mechanism of high-frequency repetitive transcranial magnetic stimulation in the treatment of upper limb bradykinesia in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Hoehn and Yahr (HY) stage 1-2
* Able to understand and cooperate with the study
* Predominantly characterized by bradykinesia
* Onset on the left side

Exclusion Criteria:

* Contraindications for TMS including DBS surgery, Ventriculoperitoneal shunt, etc
* Other neurological disorders
* Significant resting tremor, with MDS-UPDRS-III tremor score ≥3
* Resting threshold cannot be measured
* Received other TMS treatments within the last 3 months

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 2 weeks and 4 weeks
  Change in Unified Parkinson's Disease Rating Scale (MDS-UPDRS) total score of part III from Day 1 to 1 year. The part III of the MDS-UPDRS assess motor function in best on phase. The score range is 0-132, where a higher score means more severe motor impairment.

SECONDARY OUTCOMES:
cortical activation detected by fNIRS | 2 weeks and 4 weeks
  Using near-infrared brain imaging systems, have patients perform finger tapping, fist clenching, and forearm rotation movements to observe brain region activation.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China, China